CLINICAL TRIAL: NCT00380718
Title: Open-Label Single-Arm Phase IV Study of Pemetrexed in Taiwanese Patients With Advanced Non-Small Cell Lung Cancer Who Have Had Prior Chemotherapy
Brief Title: Chemotherapy for Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10720; H3E-MC-JMIC (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Results first posted 2009-10-06 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per square meter (mg/m2), intravenous (IV) in the first cycle. Acceptable toxicity* in cycle 1 determines dose increase to 1000 mg/m2 or dose decrease to 375 mg/m2 with unacceptable toxicity every 3 week in subsequent cycles till progression of disease.
  *Toxicity acceptable if none of the following toxicities recorded at any time during Cycle 1: Platelets <50 x 10^9/L; absolute neutrophil count <1.0 x 10^9/L; Stomatitis/pharyngitis/esophagitis/diarrhea Grade >2; Skin Grade >2; Serum bilirubin >3.0 x upper limit of normal (ULN); alanine aminotransferase/aspartate aminotransferase >10 x ULN; Other non-hematologic toxicities Grade >2 (except nausea, vomiting).
  Other Names: LY231514; Alimta

SUMMARY:
The purpose of this study is to assess the efficacy and toxicity of pemetrexed dosing that is tailored to individual patient tolerance in patients with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis non-small cell lung cancer (NSCLC) (Stage IIIB or IV)
* Patients' NSCLC must have progressed following one chemotherapy regimen for palliative therapy with or without subsequent targeted biological therapy
* Disease status must be that of measureable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1

Exclusion Criteria:

* Concurrent administration of any other tumor therapy
* Pregnancy or breast feeding
* Serious concomitant disorders
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-seven participants were screened; 3 did not meet inclusion/exclusion criteria and one withdrew.
Groups:
- Pemetrexed: 500 milligrams per square meter (mg/m2), intravenous (IV), every 21 days until disease progression (toxicity in cycle 1 determines dose increase to 1000 mg/m2 or dose decrease to 375 mg/m2 in subsequent cycles).
Period: Overall Study
Arm/Group | Pemetrexed
Started | 33
Received at Least One Dose of Study Drug | 33
Received Escalated Dose in Cycle 2 | 25
Completed | 15
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Death after 30-day post-therapy followup | 17

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Region of Enrollment [Number; unit: participants]
  Taiwan | 33
Disease Characteristic: Basis for Diagnosis [Number; unit: participants]
  Histopathological | 17
  Cytological | 16
Disease Characteristic: Disease Stage at Study Entry [Number; unit: participants] — Stage means how big the tumor is and how far it's spread. Stages range from 0 (the cancer has not spread beyond the inner lining of the lung) to IV (the cancer has spread to other organs of the body such as the other lung, brain, or liver).
  participants
    Stage IIIB | 3
    Stage IV | 30
Disease Characteristic: Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 9
    1 - Ambulatory, Restricted Strenuous Activity | 24
Disease Characterstic: Pathological Diagnosis Code [Number; unit: participants]
  Adenocarcinoma of Lung | 23
  Large Cell Carcinoma of Lung | 1
  Mixed Cell | 0
  Squamous Cell Carcinoma of Lung | 8
  Non-Small Cell Lung Carcinoma | 1
Race/Ethnicity [Number; unit: participants]
  East/Southeast Asian | 33
Smoking Status [Number; unit: participants]
  Ever Smoking | 20
  Never Smoking | 13
24 Hour Creatinine Clearance [Mean (Standard Deviation); unit: milliliters per minute (ml/min)] — N=32 (Data not available for 1 participant).
  milliliters per minute (ml/min) | 81.142 (24.9265)
Body Temperature [Mean (Standard Deviation); unit: degrees Celcius (°C)] | 36.25 (0.336)
Disease Characteristic: Time from Initial Diagnosis to Prior Chemotherapy Failure [Mean (Standard Deviation); unit: months] — N=25 (Data not available for 8 patients)
  months | 12.04 (23.764)
Disease Characteristic: Time from Initial Diagnosis to Study Entry [Mean (Standard Deviation); unit: months] | 11.54 (20.829)
Disease Characteristic: Time from Prior Chemotherapy Failure to Study Entry [Mean (Standard Deviation); unit: months] — N=25 (Data not available for 8 patients)
  months | 1.00 (0.486)
Heart Rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 87.5 (15.00)
Height [Mean (Standard Deviation); unit: centimeters] | 162.0 (8.59)
Homocysteine [Mean (Standard Deviation); unit: micromoles per Liter (μmol/L)] | 7.521 (2.6229)
Weight [Mean (Standard Deviation); unit: kilograms] | 63.08 (9.912)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a Complete or Partial Response (Objective Response Rate [ORR])
Description: The objective response rate (ORR) was defined as the proportion of participants who achieved a best response of either complete response (CR) or partial response (PR) (responders) based on the RECIST criteria. ORR=(CR+PR)/Number of Participants. The RECIST define when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments.
Time Frame: baseline to measured progressive disease (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until documented disease progression, or up to 18 months after enrollment)
Population: Number of participants who received at least one dose of study drug. Participants who were classified as "Unknown" were considered nonresponders rather than missing.
Measure: Mean (95% Confidence Interval); unit: proportion of responders
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
proportion of responders | 0.182 [0.07 to 0.355]

2. Secondary Outcome: Proportion of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), and Stable Disease (SD) (Disease Control Rate [DCR])
Description: DCR was defined as the proportion of best overall response of CR, PR, and SD. DCR=(CR+PR+SD)/Number of participants. Response was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
proportion of participants | 0.545 [0.364 to 0.719]

3. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death from any cause. For patients who are alive, overall survival is censored at the last follow-up visit.
Time Frame: baseline to date of death from any cause (includes post-treatment follow-up of up to 18 months post-Last Patient Entered Treatment)
Population: Number of participants who received at least one dose of study drug. Sixteen participants were censored as they were alive at the time of analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
months | 20.2 [0.7 to 32.0]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time to PFS was defined as the time from the date of enrollment to the date of the first of the following events: objective disease progression or death due to any cause. Survival time frame includes post-treatment follow-up of up to 18 months post-Last Patient Entered Treatment. Patients were censored if their disease had not progressed, treatment was discontinued due to an undocumented progression or toxicity/other reason, onset of new anti-tumor therapy or otherwise experienced death/progression after more than one missed (assessment) visit.
Time Frame: baseline to measured progressive disease or death from any cause (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until documented disease progression, or up to 18 months after enrollment)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
months | 6.9 [3.0 to 9.5]

5. Secondary Outcome: Duration of Response
Description: Duration of overall tumor response was measured from the time of first documentation of complete response or partial response (whichever status was first recorded) until the date of progression-free survival, with censoring defined as: disease had not progressed, treatment was discontinued due to undocumented progression or toxicity/other reason, onset of new anti-tumor therapy or otherwise experienced death/progression after more than one missed (assessment) visit.
Time Frame: time of response to measured progressive disease or death from any cause (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until documented disease progression, or up to 18 months after enrollment)
Population: Participants who received study drug and who had either a complete or partial response to treatment. Three participants were censored as they were alive at the time of analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 6
months | 6.6 [1.6 to 9.7]

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was define as the time from the date of enrollment to the date of the first of the following events: objective disease progression, death due to any cause, treatment discontinuation for undocumented progression, early treatment discontinuation for toxicity or other reason, or new anticancer treatment started. Time to treatment failure for participants who were still participating in the study without treatment failure at the time of analysis were treated as censored at the date of the last tumor assessment.
Time Frame: baseline to early treatment discontinuation or measured progressive disease or death from any cause (assessments every 2 cycles during therapy and 6-8 weeks during post-therapy until documented disease progression, or up to 18 months after enrollment)
Population: Number of participants who received at least one dose of study drug. One patient was censored as he/she was alive at time of analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
months | 2.9 [1.7 to 4.9]

7. Secondary Outcome: Time to Tumor Progression
Description: Time to documented tumor progression was defined as the time from the date of enrollment to the first date of documented disease progression. Time to documented disease progression was censored at the date of death for participants who had not had documented disease progression. Otherwise, the censoring rules were the same as for Progression-Free Survival.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 33
months | 6.9 [3.0 to 9.5]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=33)
Anaemia (Blood and lymphatic system disorders) | 7 (11)
Leukopenia (Blood and lymphatic system disorders) | 7 (25)
Neutropenia (Blood and lymphatic system disorders) | 5 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 7 (10)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 9 (12)
Asthenia (General disorders) | 3 (3)
Chest pain (General disorders) | 9 (10)
Fatigue (General disorders) | 11 (28)
Malaise (General disorders) | 6 (10)
Pyrexia (General disorders) | 8 (9)
Herpes virus infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
Creatinine renal clearance decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 6 (8)
Lymphocyte count decreased (Investigations) | 5 (17)
Lymphocyte percentage decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 8 (22)
White blood cell count decreased (Investigations) | 7 (20)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 4 (7)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (17)
Rash (Skin and subcutaneous tissue disorders) | 7 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days